CLINICAL TRIAL: NCT04883151
Title: The SOFUS Psychological Intervention for Families With Children in Pediatric Palliative Care - a Pilot Study
Brief Title: A Psychological Intervention for Families in Pediatric Palliative Care
Acronym: SOFUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Cancer Society (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Pernille Bidstrup, Senior researcher and group leader, Danish Cancer Society
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SOFUS
Record Dates: First submitted 2021-04-27; First posted 2021-05-12 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Distress, Emotional; Grief
Keywords: Pediatric palliative care; Family intervention; Emotion regulation; Grief intervention
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOFUS pilot program (Experimental)
  Interventions: Behavioral: SOFUS pilot program

INTERVENTIONS:
Behavioral: SOFUS pilot program — The SOFUS pilot program consists of six pre-loss sessions (Program 1) and a further six post-loss sessions (Program 2), which are delivered over a 3-month period. Each session ranges from 1-1.5 hours. Sessions 1 and 6 includes the whole family, sessions 2 and 3 focus on the parents, while sessions 4 and 5 target the children (with parents if the child is <10 years old).
  SOFUS consists of three primary components: i) strengthening COMMUNICATION between parents and children, ii) NORMALIZATION of grief processes (pre and post-lost), and iii) EMOTION REGULATION strategies targeting motivational awareness and regulatory skills in grief management (pre and post-lost).
  Families in Program 1 may be offered Program 2 if the child dies before the entire program has been delivered.

SUMMARY:
Families of children receiving pediatric palliative care report unmet needs that require support. The objective of this pilot study is to develop and evaluate a psychological intervention (SOFUS) that targets the whole family (i.e. parents, the ill child and siblings) before and after bereavement. The aim of the intervention is to improve coping skills and reduce symptoms of complicated grief, depression, anxiety and sleep disorders in families. Feasibility and acceptability of the intervention manual and study materials will be evaluated, and the preliminary efficacy of the intervention will be assessed.

DETAILED DESCRIPTION:
Having a child in palliative care is a traumatic experience and families of children receiving pediatric palliative care report unmet needs that require support. Parents who experience the death of a child often experience severe grief reactions, which may develop into long-term impaired functioning or psychiatric illness, with a detrimental impact on the whole family. Furthermore, parents and siblings of a child in palliative care may already prior to death experience grief and loss. This indicates the need for a family-based intervention that can support the family before and after the death of a child.

SOFUS is a psychological intervention for families of children receiving pediatric palliative care team. The preliminary/pilot program has been manualized and consists of a pre-loss program (Program 1) and a post-loss program (Program 2) consisting of six sessions each designed for the whole family. Sessions 1 and 6 includes the whole family, sessions 2 and 3 focus on the parents, while sessions 4 and 5 target the children (with parents if the child is under 10 years old). The six sessions range from 1 to 1.5 hours in length and are to be delivered over a 3 month period. The intervention will be carried out by trained psychologists. Feasibility and fidelity will assessed by evaluation forms filled out by the therapist after each session.

At the end of the intervention, semi-structured interviews will be carried out with each family to evaluate the components of the intervention, participant materials and assess acceptability. A semi-structured interview will also be carried out with the psychologists to evaluate the components of the intervention, the intervention manual and to assess therapist acceptability of the intervention. This pilot study will also include questionnaires for the parents assessing the outcomes of coping, anxiety, depression, sleep quality, family functioning and family caregiving burden at baseline, 3, 6 and 12 months. Age-adapted questionnaires will be given to the children to assess a subset of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Parents of a child age between 6 months and 18 years referred to the palliative team for children and adolescents
* At least one parent > 18 years
* Able to understand and speak Danish wish to participate
* Informed consent by at least one parent, and by both parents on behalf of any children participating

Exclusion Criteria:

- Any untreated psychiatric disorder or substance abuse in the family that may hinder participation in the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Satisfaction assessed by questionnaire items constructed for this study | Post-intervention (3 months)
  Measured by 9 study-specific items assessing parental satisfaction with the intervention's materials, the therapist and the intervention's focus on family/child-related factors; score range 0-27; higher scores = higher satisfaction
Satisfaction assessed by interview items constructed for this study | Post-intervention (3 months)
  Assessed through open-ended interview items evaluating the family's satisfaction with the following: 1) motivation and barriers to participation, 2) format of the intervention, 3) video and written materials of the intervention, and 4) intervention components related to the children.
Feasibility assessed by questionnaire items constructed for this study | After each session
  Measured by items assessing whether the therapist carried out each section of the manualized session and whether the time allotted was sufficient. Section scores range from 0-12, with higher scores indicating higher feasibility.
Feasibility assessed by interview items constructed for this study | Post-intervention (3 months)
  Assessed through open-ended interview items evaluating the the following: 1) recruitment procedures, 2) format of the intervention, 3) focus areas of intervention, 4) the intervention manual, and 5) the intervention materials for the families.

SECONDARY OUTCOMES:
Change in coping strategies in parents and children above 12 years | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 28-item Brief COPE Inventory consisting of 14 subscales (Self-distraction, Active coping, Denial, Substance use, Use of emotional support, Use of instrumental support, Behavioral disengagement, Venting, Positive reframing, Planning, Humor, Acceptance, Religion, and Self-blame). Scores are reported for each subscale; score range 2-8; higher scores = higher use of this specific coping strategy
Change in coping strategies in children 6-12 years old | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 15-item KidCope assessing the frequency (whether the child used the strategy) and efficacy (whether it helped) of 11 types of coping strategies (4 adaptive coping = problem solving, positive emotion regulation, cognitive restructuring, seeking social support; 7 maladaptive coping = distraction, negative emotion regulation, social withdrawal, wishful thinking, self-criticism, blaming others, resignation). Scores are reported for each coping strategy. Frequency is assessed by 1=Yes/0=No and efficacy is assessed on a scale from 0 (Not at all) to 2 (A-lot). Higher scores reflect greater use and/or perceived helpfulness of the indicated coping strategy or type of coping
Change in symptoms of grief in parents and children above 12 years | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 13-item Prolonged Grief-13 (PG-13), the pre-loss PG-13 will be used for families in Program 1. The duration and impairment items are assessed by Yes/No and score range for the remaining 11 multiple choice items = 11-44; higher scores = higher grief symptoms.
Change in symptoms of anxiety in parents and children above 12 years | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 7-item Generalized Anxiety Disorder-7 (GAD-7); range 0-21; higher scores = more symptoms
Change in symptoms of depression in parents and children above 12 | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 9-item Patient Health Questionnaire-9 (PHQ-9); range 0-27; higher scores = more symptoms
Change in symptoms of depression in children 2-5 years old | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 21-item Pediatric Emotional Distress Scale (PEDS); range 21-84; higher scores = more symptoms
Change in symptoms of depression in children 6-12 years old | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 25-item Strengths and Difficulties Questionnaire (SDQ), consisting of 5 subscales (Emotional symptoms, Conduct problems, Hyperactivity/inattention, Peer relationships problem, and Prosocial behaviour). Scores are reported for each subscale; score range 0-10. For the 4 difficulties subscales, higher scores = more difficulties; for the strength subscale, higher score = better social strength
Change in sleep quality in parents only | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the Pittsburgh Sleep Quality Index (PSQI); range 0-21; higher scores = worse sleep quality
Change in emotion regulation in parents | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 36-item Cognitive Emotion Regulation Questionnaire (CERQ) consisting of 9 subscales (Self-blame, Blaming others, Acceptance, Refocusing on planning, Positive refocusing, Rumination, Positive reappraisal, Putting into perspective, and Catastrophizing); Scores are reported by subscale; score range 4-20; higher scores = greater use of the specific cognitive strategy
Change in emotion regulation in children | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by six emotion thermometers (developed for the study) assessing guilt, jealousy, fear, happiness, sadness and anger; score range 1-10; higher scores = higher levels of emotion
Change in family functioning in parents and children above 12 years | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the Family Assessment Device (FAD) communication subscale (6 items) and general functioning subscale (12-items). Scores are reported by subscale; score range 1-4; higher scores = better family functioning
Change in family caregiving burden in parents only | Between baseline and 3 months, 6 months, 12 months, respectively
  Measured by the 25-item Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC) consisting of 4 subscales (caregiver strain, positive caregiving appraisals, caregiver distress, and family well-being. Scores are reported by subscale; score range 1-5; higher scores = higher level on the specific subscale measure.

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Bidstrup, PhD, Principal Investigator — Danish Cancer Society Research Center
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No